CLINICAL TRIAL: NCT06859268
Title: A Phase 3b, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate Retatrutide Treatment in the Maintenance of Weight Reduction in Individuals With Obesity
Brief Title: A Study of Retatrutide (LY3437943) in the Maintenance of Weight Reduction in Individuals With Obesity
Acronym: TRIUMPH-6
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27268; J1I-MC-GZQB (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-02-28; First posted 2025-03-05 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — retatrutide

STUDY DESIGN:
Intervention Model Description: Phase 3b
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Retatrutide Dose 1 (Experimental): Participants will receive retatrutide dose 1 administered subcutaneously (SC) for 116 weeks
  Interventions: Drug: Retatrutide
- Retatrutide Dose 1 to Retatrutide Dose 2 (Experimental): Participants will receive retatrutide dose 1 administered SC for 80 weeks, then retatrutide dose 2 administered SC for an additional 36 weeks
  Interventions: Drug: Retatrutide
- Retatrutide Dose 1 to Placebo (Placebo Comparator): Participants will receive retatrutide dose 1 administered SC for 80 weeks, then placebo administered SC for an additional 36 weeks
  Interventions: Drug: Retatrutide; Drug: Placebo

INTERVENTIONS:
Drug: Retatrutide — Administered SC
  Other Names: LY3437943
Drug: Placebo — Administered SC
  Arms: Retatrutide Dose 1 to Placebo

SUMMARY:
This is a study of retatrutide in participants with obesity. The main purpose is to learn more about how retatrutide maintains body weight loss. The study will have two treatment phases: an 80 week lead-in phase in which all participants will take retatrutide dose 1 and a 36 week randomized, double-blinded phase in which participants will either take retatrutide dose 1, retatrutide dose 2, or switch to placebo. Participation in the study will last around 125 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have obesity and a history of at least one self-reported unsuccessful dietary effort to reduce body weight

Exclusion Criteria:

* Have a self-reported change in body weight >5 kilograms (kg) (11 pounds) within 90 days before screening
* Have a prior or planned surgical treatment for obesity
* Have a prior or planned endoscopic procedure and/or device-based therapy for obesity
* Have Type 1 Diabetes, Type 2 Diabetes, or any other type of diabetes
* Have a family or personal history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN-2)
* Have had within the past 90 days before screening:

  * acute myocardial infarction
  * cerebrovascular accident (stroke)
  * hospitalization for unstable angina, or
  * hospitalization due to congestive heart failure
* Have New York Heart Association Functional Classification Class IV congestive heart failure
* Have a history of chronic or acute pancreatitis
* Have taken weight loss drugs, including over-the-counter medications, within 90 days prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 643 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Percent Change from Baseline in Body Weight | Week 0, Week 116

SECONDARY OUTCOMES:
Change from Baseline in Waist Circumference | Week 0, Week 116
Percentage of Body Weight Reduction Achieved at Week 80 that is Maintained at Week 116 | Week 0, Week 80, Week 116
Change from Baseline in Impact of Weight on Quality of Life-Lite Clinical Trials Version (IWQOL-Lite-CT) | Week 0, Week 116

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (53):
- United States (33):
  - Southern California Clinical Research, Santa Ana, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - CMR of Greater New Haven, LLC, Hamden, Connecticut
  - ALL Medical Research, LLC, Cooper City, Florida
  - Florida International Medical Research, Coral Gables, Florida
  - Renstar Medical Research, Ocala, Florida
  - Charter Research - Winter Park, Orlando, Florida
  - Metabolic Research Institute, Inc., West Palm Beach, Florida
  - Kubost Clinical Research - Marietta, Marietta, Georgia
  - North Georgia Clinical Research, Woodstock, Georgia
  - Pacific Diabetes & Endocrine Center, Honolulu, Hawaii
  - Alliance for Multispecialty Research, LLC, Oak Brook, Illinois
  - Springfield Clinic Main Campus, Springfield, Illinois
  - Alliance for Multispecialty Research, LLC, Lexington, Kentucky
  - L-MARC Research Center, Louisville, Kentucky
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Care Access - Lake Charles (Bayou Pines), Lake Charles, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Alliance for Multispecialty Research, LLC, Kansas City, Missouri
  - Vector Clinical Trials, Las Vegas, Nevada
  - Dent Neurosciences Research Center, Inc, Amherst, New York
  - Carteret Medical Group, Morehead City, North Carolina
  - Care Access - Raleigh, Raleigh, North Carolina
  - Tekton Research, LLC., Moore, Oklahoma
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - Care Access - Rapid City, Rapid City, South Dakota
  - Alliance for Multispecialty Research, LLC, Knoxville, Tennessee
  - Care Access - Houston, Houston, Texas
  - Southern Endocrinology Associates, Mesquite, Texas
  - Sleep Therapy Research Center, San Antonio, Texas
  - National Clinical Research, Inc, Richmond, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Central Washington Health Services Association d/b/a Confluence Health, Wenatchee, Washington
- Canada (8):
  - Aggarwal and Associates Limited, Brampton
  - Circulate Cardiac & Vascular Centre, Burlington
  - Med Trust Research, Courtice
  - Winterberry Research Inc., Hamilton
  - Centre de Medecine Metabolique de Lanaudiere (CMML), Terrebonne
  - Care Access - Thunder Bay - Barton Street, Thunder Bay
  - Maple Leaf Research, Toronto
  - C.I.C. Mauricie inc., Trois-Rivières
- United Kingdom (12):
  - FutureMeds - Birmingham, Birmingham
  - Oakenhurst Medical Practice, Blackburn
  - Layton Medical Centre, Blackpool
  - Bradford on Avon Health Centre, Bradford-on-Avon
  - FutureMeds - Liverpool, Bromborough
  - Cheadle Community Hospital, Cheadle
  - HMC Health Group - Meadows Centre for Health, Hounslow
  - St Bartholomew's Medical Centre, Oxford
  - Atlantic Medical, Penzance
  - The Adam Practice, Poole
  - Woodstock Bower Surgery, Rotherham
  - Rame Group Practice, Torpoint

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of Retatrutide (LY3437943) in the Maintenance of Weight Reduction in Individuals with Obesity (TRIUMPH-6) — https://trials.lilly.com/en-US/trial/580035